CLINICAL TRIAL: NCT03726957
Title: Exploring Respiratory Health Outcomes From Sustained Use of Efficient Cookstoves
Acronym: STAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: Washington University School of Medicine (Other); Sri Ramachandra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1R21ES021585-01A1 (NIH)
Record Dates: First submitted 2018-10-17; First posted 2018-11-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Intervention Model Description: The investigators adopted a cluster randomized controlled trial with village as the unit of randomization. Villages were randomized to have participating households assigned to either a traditional biomass burning cookstove (control group) or to an improved cookstove (intervention group). A household that was willing to participate was considered eligible: 1) if it had a traditional wood burning cookstove; and 2) if the household included at least one child between the ages of 8-15. If a household had more than one child within the target age range, the oldest child within the age range was selected for study. Study participants within each household were the mother and the selected child.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention arm included households which received improved cookstoves
  Interventions: Behavioral: Improved Cookstoves
- Control group (No Intervention): The control group included households, which did not receive improved cookstoves, and cooked in their usual traditional cookstoves.

INTERVENTIONS:
Behavioral: Improved Cookstoves — Villages were randomized to have participating households assigned to either a traditional biomass burning cookstove or to an improved cookstove. Once the participating villages had been selected, the investigators used their list of eligible households within each village to randomly order these households. Within each village, the investigators then approached the eligible households in the order that had been randomly chosen and continued that process until four households within each village had agreed to participate. The selection of villages and households preceded randomization and was pursued with the clear understanding that group assignment would be random, and that participation reflected a willingness to be randomized to either study group.
  Arms: Intervention group

SUMMARY:
Household air pollution (HAP) is a leading risk factor for global burden of disease. Resource-constrained communities of the world especially women and children are significantly impacted by this challenge. To address household air pollution, cleaner and more efficient improved cookstoves (ICS) have been disseminated to low resource communities. Although there has been initial uptake of these stoves, sustained use has been inconsistent adding to the challenge of household air pollution. There is limited understanding at the intersections of social, ecological, and technical determinants of sustained use of ICS, and how is sustained use of ICS associated with exposure and health outcomes in poor communities.

The overarching goal of this exploratory study is to initiate a comprehensive research program that will facilitate the use of ICS and investigate whether they render significant health benefits among rural Indian households.

The investigators installed ICS (model: Eco-Chulla XXL) in select households that primarily use biomass for cooking, and evaluate the intervention based on three specific aims:

1. To generate preliminary emissions data [particulate matter - mass and surface area based, carbon monoxide (CO)] from ICS and its effect on respiratory health outcomes that will facilitate the development of a pivotal clean cookstove intervention
2. To generate effect size data that establish the feasibility and inform the sample size of a pivotal trial whose primary objective will be sustained improvements in the respiratory health of women and children in rural India
3. To evaluate factors which enable and hinder the sustained use of clean cookstove technologies by the rural poor in India so that the investigators can develop a more refined pivotal intervention focused on improving respiratory health

DETAILED DESCRIPTION:
In this study, the investigators undertake a 12-month cluster randomized trial in 96 households in the rural areas of Andhra Pradesh and Karnataka states of India. The investigators enrolled women (primary cook) and one child (age 8-15) in each of these 96 households. The investigators compare the effect of traditional wood burning stoves (the control condition) to that of improved wood burning stoves on the respiratory health of women and children, and also undertake community-based system dynamics modeling to delineate the feedback mechanisms involved in sustained use or abandonment of improved cookstoves. The study and research program are aligned with recent international attention to explore determinants impacting the sustained use of cleaner cooking systems in poor communities of the world. Thus, in achieving the aims of this R21, the investigators will then have: 1) necessary preliminary data; 2) pre-emptive strategies for most of these unanticipated but preventable challenges. The investigators will leverage these insights to proceed with a larger scale intervention: 1) to examine the effect of sustained use of cleaner cooking systems and respiratory health outcomes in women and children due to reduced HAP in rural India; 2) to explore barriers and enablers of implementation of cleaner cooking systems in multiple resource poor settings. Numerous studies have shown that sustained and exclusive use of cleaner cooking systems irrespective of their types have been a challenge. Lukewarm sustenance of cleaner cooking systems in poor households stems from a limited understanding on the grounds of social, technical, economic, and ecological intersections of energy security. The investigators intend to address this gap by using a trans-disciplinary approach to contribute to our understanding of factors that influence the implementation of cleaner cooking systems for rural poor in India.

ELIGIBILITY:
Inclusion criteria:

* The household had a traditional wood burning cookstove and had at least one woman (primary cook) at least the age of 18, and one child between age 8-15 (both included).
* If a household had more than one child within the target age range, the oldest child within the age range was selected for study.

Exclusion criteria:

• Both the woman and the child could not successfully undertake spirometry.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-12-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume 1 (FEV1) | 12 months
  The investigators used Koko spirometer to measure the forced expiratory volume in 1 second (FEV1).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel S, Leavey A, Sheshadri A, Kumar P, Kandikuppa S, Tarsi J, Mukhopadhyay K, Johnson P, Balakrishnan K, Schechtman KB, Castro M, Yadama G, Biswas P. Associations between household air pollution and reduced lung function in women and children in rural southern India. J Appl Toxicol. 2018 Nov;38(11):1405-1415. doi: 10.1002/jat.3659. Epub 2018 Jul 25. PMID 30047157